CLINICAL TRIAL: NCT05270668
Title: A Double Blind, Randomized, Placebo-Controlled Study to Evaluate the Efficacy and Safety of MK-7240/PRA023 in Subjects With Systemic Sclerosis Associated With Interstitial Lung Disease (SSc-ILD)
Brief Title: Phase 2 Safety and Efficacy Study of Tulisokibart (MK-7240/PRA023) in Subjects With Systemic Sclerosis Associated With Interstitial Lung Disease (SSc-ILD) (MK-7240-007)
Acronym: ATHENA-SSc-ILD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Prometheus Biosciences, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7240-007; PR200-104 (Other: PrometheusBio); MK-7240-007 (Other: MSD); 2023-509743-27-00 (Registry Identifier: EU CT); U1111-1309-6150 (Registry Identifier: UTN); 2021-005206-10 (EudraCT Number)
Record Dates: First submitted 2022-02-27; First posted 2022-03-08 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-07

CONDITIONS: Diffuse Cutaneous Systemic Sclerosis; Interstitial Lung Disease
Keywords: ATHENA SSc-ILD; ATHENA; Diffuse Cutaneous Scleroderma; Interstitial Lung Disease
MeSH Terms: conditions — Scleroderma, Diffuse; Lung Diseases, Interstitial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Tulisokibart (Experimental): Tulisokibart IV administered by IV infusion
  Interventions: Drug: Tulisokibart; Diagnostic Test: Companion diagnostic ( CDx)
- Placebo (Placebo Comparator): Placebo administered by IV infusion
  Interventions: Diagnostic Test: Companion diagnostic ( CDx); Drug: Placebo

INTERVENTIONS:
Drug: Tulisokibart — Tulisokibart administered at timepoints as directed by the protocol
  Other Names: PRA023; MK-7240
  Arms: Tulisokibart
Diagnostic Test: Companion diagnostic ( CDx) — CDx+ or CDx-
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of tulisokibart in participants with SSc-ILD.

ELIGIBILITY:
Inclusion Criteria:

* Has confirmed diagnosis of systemic sclerosis with onset of disease ≤ 5 years ago.
* Has diffuse cutaneous scleroderma
* Has systemic sclerosis related interstitial lung disease confirmed by HRCT
* FVC ≥ 45% of predicted normal
* Diffusing capacity of lung for carbon monoxide (DLCO)≥ 45% of predicted normal
* If on background therapy, meets stable dosing requirements for nintedanib, mycophenolate mofetil (MMF), methotrexate (MTX) OR azathioprine, and corticosteroids
* Women of childbearing potential are eligible to participate if not pregnant or breastfeeding and either willing to use an acceptable contraceptive method or sexually abstinent
* Able to provide written informed consent and understand and comply with the requirements of the study

Exclusion Criteria:

* Has an airway obstruction per pulmonary function test (PFT) or clinically significant pulmonary arterial hypertension
* Has current clinical diagnosis of another inflammatory connective tissue disease
* Has any active infections, a serious infection within the past 3 months, or chronic bacterial infection
* Is a current smoker or smoking within 6 months of screening
* Has any concomitant medical conditions that, in the opinion of the investigator, might place them in unacceptable risk for participation in the study
* Meets the protocol criteria for important laboratory exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who Experience an Adverse Event (AE) | Up to Week 50
  An AE is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. The number of participants who experience an AE will be reported.
Number of Participants who Experience a Serious Adverse Event (SAE) | Up to Week 50
  An AE is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. The number of participants who experience an SAE will be reported.
Number of Participants who Discontinue due to an AE | Up to Week 50
  An AE is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. The number of participants who discontinue due to an AE will be reported.
Change from Baseline in the Annual Rate of Change in Forced Vital Capacity (FVC) at Week 50 | Baseline and up to Week 50
  FVC, as measured in milliliters by spirometry, is the amount of air forcibly exhaled from the lungs after taking the deepest breath possible.

SECONDARY OUTCOMES:
Change from Baseline in FVC at Week 50 | Baseline and Week 50
  FVC, as measured in milliliters by spirometry, is the amount of air forcibly exhaled from the lungs after taking the deepest breath possible.
Change from Baseline in High-Resolution Computer Tomography (HRCT) Quantitative Interstitial Lung Disease - Whole Lung (QILD-WL) at Week 50 | Baseline and Week 50
  QILD-WL will be measured as percent lung involvement using HRCT.
Percentage of Participants with an Improvement in the Revised Composite Response Index in Systemic Sclerosis (CRISS) Score at Week 50 | Baseline and Week 50
  The Revised CRISS is a two-step process designed to evaluate the likelihood of improvement in early SSc. The first step assesses worsening or incident cases of internal organ involvement (scleroderma renal crisis, pulmonary arterial hypertension, congestive heart failure, ILD, severe gastrointestinal dysmotility requiring parenteral or enteral nutrition, and digital ischemia requiring hospitalization, gangrene, or amputation). The second step assesses changes from baseline in five core set measures: modified Rodnan skin score (mRSS), percent predicted forced vital capacity (FVC%), health assessment questionnaire-disability index (HAQ-DI), patient (PGA), and physician (PhGA) global assessments.
Change from Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 50 | Baseline and Week 50
  HAQ is an instrument to assess physical function. It consists of 20 questions, covering eight types of activities. For each question, scores range from 0 to 3 (0 = without any difficulty; 1 = with some difficulty; 2 = with much difficulty or with assistance; 3 = unable to do). HAQ Disability Index (HAQ-DI) score is the average of the highest score in each of the eight categories.
Change from Baseline in Living with Pulmonary Fibrosis (L-PF) Quality of Life (QoL) Outcome at Week 50 | Baseline and Week 50
  The L-PF is a questionnaire designed to assess the quality of life of patients with pulmonary fibrosis. It contains 44 questions (items) split into two modules, 23 which assess symptoms (including shortness of breath, cough, and fatigue) and 21 which assess impacts to quality of life. Individual items are scored on a 5-point scale (0 = Not at All to 4 = Extremely). Overall scores range from 0 to 100 with higher scores indicating a greater impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Prometheus Biosciences, Study Director — Clinical Trials Call Center
Locations (95):
- United States (20):
  - Mayo Clinic - Scottsdale ( Site 4014), Phoenix, Arizona
  - Pacific Arthritis Care Center ( Site 4008), Los Angeles, California
  - Cedars Sinai Medical Center ( Site 4010), Los Angeles, California
  - UCLA School of Medicine ( Site 4006), Los Angeles, California
  - Stanford Health Care ( Site 4009), Palo Alto, California
  - National Jewish Health Medical Center ( Site 4015), Denver, Colorado
  - Yale University ( Site 4017), New Haven, Connecticut
  - MedStar Georgetown University Hospital ( Site 4005), Washington D.C., District of Columbia
  - Johns Hopkins Asthma and Allergy Center [Baltimore, MD] ( Site 4018), Baltimore, Maryland
  - Massachusetts General Hospital ( Site 4003), Boston, Massachusetts
  - Boston University School of Medicine ( Site 4021), Boston, Massachusetts
  - University of Michigan Hospital ( Site 4001), Ann Arbor, Michigan
  - Rutgers Robert Wood Johnson Medical School ( Site 4013), New Brunswick, New Jersey
  - Hospital For Special Surgery ( Site 4020), New York, New York
  - Cleveland Clinic Foundation ( Site 4019), Cleveland, Ohio
  - University of Toledo Medical Center ( Site 4002), Toledo, Ohio
  - University of Pittsburgh Medical Center ( Site 4016), Pittsburgh, Pennsylvania
  - Medical University of South Carolina - PPDS ( Site 4004), Charleston, South Carolina
  - UT Physicians Rheumatology ( Site 4007), Houston, Texas
  - Froedtert and Medical College of Wisconsin ( Site 4012), Milwaukee, Wisconsin
- Argentina (4):
  - Consultorios Médicos Dr. Doreski ( Site 4800), CABA, Buenos Aires
  - Clínica Privada Independencia ( Site 4802), Munro, Buenos Aires
  - Centro de Investigación Instituto Médico Río Cuarto ( Site 4801), Río Cuarto, Córdoba Province
  - Instituto Medico de la Fundacion Estudios Clinicos ( Site 4803), Rosario, Santa Fe Province
- Australia (2):
  - Royal Adelaide Hospital ( Site 4050), Adelaide, South Australia
  - St Vincents Hospital Melbourne ( Site 4051), Melbourne, Victoria
- Belgium (3):
  - UZ Gent ( Site 4401), Ghent, Oost-Vlaanderen
  - UZ Leuven ( Site 4402), Leuven, Vlaams-Brabant
  - CHU de Liege ( Site 4400), Liège, Wallonne, Region
- Canada (3):
  - University Of Alberta Hospital ( Site 4702), Edmonton, Alberta
  - St. Joseph's Health Care London ( Site 4701), London, Ontario
  - Mount Sinai Hospital [Toronto, Canada] ( Site 4700), Toronto, Ontario
- Chile (6):
  - BIOCINETIC Ltda ( Site 4854), Santiago, Region M. de Santiago
  - Centro de Investigacion Clinica UC CICUC ( Site 4855), Santiago, Region M. de Santiago
  - Centro Internacional de Estudios Clinicos CIEC ( Site 4851), Santiago, Region M. de Santiago
  - Clinica Dermacross ( Site 4853), Vitacura, Region M. de Santiago
  - Centro de especialidades médicas Vanguardia ( Site 4850), Temuco, Región de la Araucanía
  - ONCOCENTRO APYS ( Site 4852), Viña del Mar, Región de Valparaíso
- France (3):
  - CHU de Bordeaux. Hopital Pellegrin ( Site 4202), Bordeaux, Nord
  - Hôpital Claude Huriez ( Site 4200), Lille, Nord
  - Hopital Cochin ( Site 4203), Paris
- Germany (4):
  - Universitaetsklinikum Freiburg ( Site 4152), Freiburg im Breisgau, Baden-Wurttemberg
  - Kerckhoff-Klinik-Forschungs-GmbH ( Site 4153), Bad Nauheim, Hesse
  - Rheumazentrum am Krankenhaus Bad Doberan ( Site 4150), Hohenfelde B Bad Doberan, Mecklenburg-Vorpommern
  - Universitaetsklinikum Koeln ( Site 4151), Cologne, North Rhine-Westphalia
- Hungary (4):
  - Pecsi Tudomanyegyetem AOK ( Site 4250), Pécs, Baranya
  - Budai Irgalmasrendi Korhaz ( Site 4252), Budapest
  - Del-pesti Centrumkorhaz Orszagos Hematologiai es Infektologiai Intezet ( Site 4253), Budapest
  - Debreceni Egyetem Klinikai Kozpont ( Site 4251), Debrecen
- Israel (6):
  - Rambam Medical Center ( Site 4601), Haifa
  - Meir Medical Center. ( Site 4604), Kfar Saba
  - Galilee Medical Center ( Site 4602), Nahariya
  - Rabin Medical Center ( Site 4603), Petach Tikvah
  - Sheba Medical Center ( Site 4605), Ramat Gan
  - Tel Aviv Sourasky Medical Center ( Site 4606), Tel Aviv
- Italy (8):
  - A.O.U. Citta della Salute e della Scienza di Torino ( Site 4304), Turin, Piedmont
  - Azienda Ospedaliera Universitaria Careggi ( Site 4301), Florence
  - Ospedale Policlinico San Martino ( Site 4305), Genova
  - IRCCS Osp. Maggiore Policlinico ( Site 4306), Milan
  - Ospedale San Raffaele di Milano ( Site 4307), Milan
  - Fondazione IRCCS Policlinico San Matteo ( Site 4303), Pavia
  - Arcispedale Santa Maria Nuova ( Site 4300), Reggio Emilia
  - Azienda Policlinico Umberto I ( Site 4302), Roma
- Mexico (2):
  - PanAmerican Clinical Research - Guadalajara ( Site 4900), Guadalajara, Jalisco
  - Centro de Investigación y Tratamiento Reumatológico S.C ( Site 4902), Mexico City, Mexico City
- Radboud University Medical Center ( Site 4650), Nijmegen, Gelderland, Netherlands
- Oslo Universitetssykehus HF. Rikshospitalet ( Site 4350), Oslo, Norway
- Instituto de Ginecologia y Reproduccion ( Site 4952), Lima, Peru
- Poland (7):
  - Twoja Przychodnia Poznanskie Centrum Medyczne ( Site 4452), Poznan, Greater Poland Voivodeship
  - Narodowy Instytut Geriatrii Reumatologii i Rehabilitacji im.Prof. El. Reicher-ul.Spartanska 1 ( Site, Warszawa, Greater Poland Voivodeship
  - Szpital Uniwersytecki nr 2 im. dr Jana Biziela w Bydgoszczy ( Site 4454), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Centrum Medyczne Oporow ( Site 4455), Wroclaw, Lower Silesian Voivodeship
  - Centrum Medyczne Reuma Park NZOZ ( Site 4450), Warsaw, Masovian Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku - Marii Sklodowskiej-Curie 24A ( Site 4451), Bialystok, Podlaskie Voivodeship
  - Szpital Specjalistyczny nr 1 w Bytomiu ( Site 4453), Bytom, Silesian Voivodeship
- Spain (9):
  - HOSPITAL CLÍNIC DE BARCELONA ( Site 4105), Barcelona, Catalonia
  - Hospital Universitario 12 de Octubre ( Site 4106), Madrid, Madrid, Comunidad de
  - Hospital Central de Asturias ( Site 4109), Oviedo, Principality of Asturias
  - Hospital Universitario Vall d'Hebron - PPDS ( Site 4107), Barcelona
  - Hospital Santa Creu i Sant Pau ( Site 4102), Barcelona
  - Hospital Universitario Ramon y Cajal ( Site 4101), Madrid
  - Hospital Regional Universitario de Malaga ( Site 4104), Málaga
  - Hospital Universitario Doctor Peset ( Site 4103), Valencia
  - Hospital Clinico Universitario Lozano Blesa ( Site 4100), Zaragoza
- Switzerland (4):
  - Inselspital Bern ( Site 4502), Bern, Canton of Bern
  - Kantonsspital St. Gallen ( Site 4501), Sankt Gallen, Canton of St. Gallen
  - Hopitaux Universitaires de Geneve HUG ( Site 4503), Geneva
  - Universitaetsspital Zuerich ( Site 4500), Zurich
- Ukraine (5):
  - Kyiv City Clinical Hospital # 3 ( Site 4754), Kyiv, Kyivska Oblast
  - ME "Ternopil Regional Clinical Hospital of Ternopil Regional Council" ( Site 4750), Ternopil, Ternopil Oblast
  - Vinnytsia Nat Med University n.a.M.Pyrogov,City Clinical Hospital #1 ( Site 4751), Vinnytsia, Vinnytsia Oblast
  - Medical Center OK!Clinic+LLC International Institute of Clinical Research ( Site 4753), Kyiv
  - Institute of Rheumatology LLC ( Site 4752), Kyiv
- United Kingdom (2):
  - Royal Free Hospital ( Site 4550), London, London, City of
  - Chapel Allerton Hospital ( Site 4551), Leeds

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26198&tenant=MT_MSD_9011